CLINICAL TRIAL: NCT06352424
Title: A Single-dose, Randomized, Placebo-controlled Phase I Study on the Effects of a Subcutaneous Dose of BI 1820237 and BI 456906, and Combination Thereof on Functional MRI Measurements in Otherwise Healthy Male and Female Individuals With Obesity/Overweight (Single-blind, Cross-over Design)
Brief Title: A Study in People With Overweight or Obesity to Test How BI 1820237, BI 456906, or a Combination of Both Affects Brain Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1458-0006; 2023-506233-30-01 (Registry Identifier: CTIS (EU)); U1111-1293-4672 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A-B-C-D (Experimental): * A: Treatment Test 1 (T1): BI 1820237 + Placebo for BI 456906
  * B: Treatment Test 2 (T2): BI 456906 + Placebo for BI 1820237
  * C: Treatment Test 3 (T3): BI 1820237 + BI 456906
  * D: Treatment Reference (R1, R2): Placebo for BI 1820237 + Placebo for BI 456906
  Interventions: Drug: BI 456906; Drug: BI 1820237; Drug: Placebo for BI 1820237; Drug: Placebo for BI 456906
- B-D-A-C (Experimental)
  Interventions: Drug: BI 456906; Drug: BI 1820237; Drug: Placebo for BI 1820237; Drug: Placebo for BI 456906
- C-A-D-B (Experimental)
  Interventions: Drug: BI 456906; Drug: BI 1820237; Drug: Placebo for BI 1820237; Drug: Placebo for BI 456906
- D-C-B-A (Experimental)
  Interventions: Drug: BI 456906; Drug: BI 1820237; Drug: Placebo for BI 1820237; Drug: Placebo for BI 456906

INTERVENTIONS:
Drug: BI 456906 — BI 456906
Drug: BI 1820237 — BI 1820237
Drug: Placebo for BI 1820237 — Placebo for BI 1820237
Drug: Placebo for BI 456906 — Placebo for BI 456906

SUMMARY:
The main objective of this trial is to investigate the effect of BI 1820237 alone, BI 456906 alone, combination of BI 1820237 and BI 456906 versus placebo on brain activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with obesity/overweight (otherwise healthy) according to the assessment of the Investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 40 to 60 years (inclusive)
3. Body mass index (BMI) of 27.0 to 40.0 kg/m2 (inclusive). Overweight/obesity should be due to excess adipose tissue, as judged by the Investigator
4. Body weight greater than or equal to 75 kg
5. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
6. Male trial participants without need for contraception
7. Female trial participants, only if any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 2 months after last administration of trial medication are met:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (intravaginal or transdermal)
   * Bilateral tubal occlusion
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm according to verbal confirmation of female participant) and provided that partner is the sole sexual partner of the trial participant
   * Abstention from male-female sex. This is defined as being in line with the preferred and usual lifestyle of the patient. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods; declaration of abstinence for the duration of exposure to study drug, and withdrawal are not acceptable.

Or female subject meets any of the following criteria:

* Permanent sterilisation by hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy
* Woman is postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm and assessed as clinically relevant by the investigator
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signal changes following treatment with single dose of BI 1820237 alone, BI 456906 alone, and combination of BI 1820237 + BI 456906 versus placebo | 32 days plus up to 8 weeks wash-out for each sequence, up to 51 weeks
  * in the fasted state in response to food visual stimuli and nutrient-specific food preference
  * assessed by task based functional magnetic resonance imaging (fMRI) in the whole brain

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com